CLINICAL TRIAL: NCT05599802
Title: An Open-Label, Phase 1 Clinical Study to Determine the Safety and Preliminary Immunogenicity of SARS-CoV-2 Variant mRNA Vaccine (LVRNA010) in Healthy Participants Aged 18 Years and Older
Brief Title: Clinical Study of SARS-CoV-2 Variant mRNA Vaccine in Healthy Participants
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: AIM Vaccine Co., Ltd. (Industry)
Collaborators: Ningbo Rongan Biological Pharmaceutical Co., Ltd. (Industry); LiveRNA Therapeutics Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LVRNA010-I-01
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-09

CONDITIONS: SARS-CoV-2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 1A: 50μg SARS-CoV-2 variant mRNA vaccine (Experimental): Participants who have not received any COVID-19 vaccines will vaccinate two doses of study vaccine with 28 days apart.
  Interventions: Biological: SARS-CoV-2 variant mRNA vaccine low dose
- 1B: 100μg SARS-CoV-2 variant mRNA vaccine (Experimental): Participants who have not received any COVID-19 vaccines will vaccinate two doses of study vaccine with 28 days apart.
  Interventions: Biological: SARS-CoV-2 variant mRNA vaccine high dose
- 2A: 50μg SARS-CoV-2 variant mRNA vaccine (Experimental): Participants who have received 2 dose of COVID-19 inactivated vaccines will vaccinate 1 doses of study vaccine.
  Interventions: Biological: SARS-CoV-2 variant mRNA vaccine low dose
- 2B: 100μg SARS-CoV-2 variant mRNA vaccine (Experimental): Participants who have received 2 dose of COVID-19 inactivated vaccines will vaccinate 1 doses of study vaccine.
  Interventions: Biological: SARS-CoV-2 variant mRNA vaccine high dose
- 3A: 50μg SARS-CoV-2 variant mRNA vaccine (Experimental): Participants who have received 2 dose of COVID-19 mRNA vaccines will vaccinate 1 doses of study vaccine.
  Interventions: Biological: SARS-CoV-2 variant mRNA vaccine low dose
- 3B: 100μg SARS-CoV-2 variant mRNA vaccine (Experimental): Participants who have received 2 dose of COVID-19 mRNA vaccines will vaccinate 1 doses of study vaccine.
  Interventions: Biological: SARS-CoV-2 variant mRNA vaccine high dose

INTERVENTIONS:
Biological: SARS-CoV-2 variant mRNA vaccine low dose — 50μg/dose
  Arms: 1A: 50μg SARS-CoV-2 variant mRNA vaccine; 2A: 50μg SARS-CoV-2 variant mRNA vaccine; 3A: 50μg SARS-CoV-2 variant mRNA vaccine
Biological: SARS-CoV-2 variant mRNA vaccine high dose — 100μg/dose
  Arms: 1B: 100μg SARS-CoV-2 variant mRNA vaccine; 2B: 100μg SARS-CoV-2 variant mRNA vaccine; 3B: 100μg SARS-CoV-2 variant mRNA vaccine

SUMMARY:
An Open-Label, Phase 1 Clinical Study to Determine the Safety and Preliminary Immunogenicity of SARS-CoV-2 Variant mRNA Vaccine (LVRNA010)

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older.
* Understand the content of the ICF, and voluntarily sign the ICF (If the participant is unable to sign the ICF on his/her own due to illiteracy, an impartial witness is needed).
* Participants who are willing and able to comply with all scheduled visits, vaccination plan, laboratory tests, lifestyle considerations, and other study procedures.
* Female participants of childbearing potential or partners of male participants: voluntarily agree to use effective contraception with their partners prior to the (1st dose of) vaccination and must agree to continue such precautions during the study until 3 months after (full) vaccination.[Effective contraception includes oral contraceptives, injectable or implantable contraception, extended-release topical contraceptives, hormonal patches, intrauterine devices(IUDs), sterilization, abstinence, condoms (for male), diaphragms, cervical caps, etc.].
* For female participants: without childbearing potential (amenorrhea for at least 1 year or documented surgical sterilization) or have used effective contraception with a negative pregnancy test before (each dose of) vaccination in this study.
* On the day of vaccination and 24 hours prior to (each dose of) vaccination, axillary temperatures<37.3℃/99.1°F.
* Healthy participants or participants with mild underlying disease [in a stable state without exacerbation (no admission to hospital or no major adjustment to treatment regimen, etc.) for at least 3 months prior to enrollment in this study].
* (For group 2 and group 3 only) Participants who have received full primary vaccination of licensed SARS-CoV-2 vaccine (3-8 weeks between 2 doses of COVID-19 inactivated vaccine or 2 doses of COVID-19 mRNA vaccine) and whose last dose was given >6 mony
* (For group 1 only) Not have received any COVID-19 vaccine prior to enrollment.

Exclusion Criteria:

* Any screening hematology and/or blood biochemistry laboratory value that meets the definition of a ≥Grade 1 abnormality,
* (For group 1 only) Confirmed SARS-CoV-2 diagnosis within 1 years before screening visit.
* History of Severe Acute Respiratory Syndrome (SARS), Middle East Respiratory Syndrome (MERS), or other coronavirus infections.
* Receipt of medications intended to treat COVID-19 with 1 year.
* History of server adverse reaction associated with a vaccine or drug and/or severe allergic reaction (e.g., anaphylaxis) to any component of the study intervention(s).
* SARS-CoV-2 RT-PCR positive nasopharyngeal/oropharyngeal swab specimens at screening.
* Positive HIV test at screening.
* A history or family history of convulsions, epilepsy, encephalopathy and psychosis.
* Malignant tumors in the active phase, malignant tumors not receiving adequate treatment, malignant tumors at potential risk of recurrence during the study period.
* Asplenia of functional asplenia, complete or partial splenectomy from any cause.
* Individuals who receive treatment with radiotherapy or immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids (if systemic corticosteroids are administered for≥14 days at a dose of ≥20 mg/day of prednisone or equivalent), e.g., for cancer or an autoimmune disease, or planned receipt throughout the study. Inhaled/nebulized, intra-articular, epidural, or topical (skin or eyes) corticosteroids are permitted.
* Any other licensed vaccines given within 28 days prior to the investigational vaccination, or planned administration of vaccine(s) within 28 days after (full) vaccination.
* Receipt of blood/plasma products, immunoglobulin, or monoclonal antibodies, form 60 days before vaccine administration, or receipt of any passive antibody therapy specific to COVID-19, from 90 days before vaccine administration, or planned receipt throughout the study.
* Blood donation or blood loss ≥450ml within 1 month prior to enrollment or planned to donate blood during the study period.
* Participation in other studies involving study intervention within 28 days prior to study entry, and/or during the study.
* Women who are pregnant or breastfeeding.
* Participants deemed unsuitable for participation in this study based on the investigator's assessment.
* (For group 1 only: Criteria for delay of 2nd dose of vaccination) Fever within 24 hours prior to the 2nd dose of vaccination (axillary body temperature ≥37.3℃/99.1°F).
* (For group 1 only: Criteria for delay of 2nd dose of vaccination) During treatment/recovery from illness.
* (For group 1 only: Criteria for delay of 2nd dose of vaccination) Other conditions considered by the investigator to be unsuitable for vaccination.
* (For group 1 only: Criteria for termination of 2nd dose of vaccination) Participants with a positive urine pregnancy or blood pregnancy test (women of childbearing age only).
* (For group 1 only: Criteria for termination of 2nd dose of vaccination) Serious allergic reactions or serious adverse events related to vaccination (as assessed by the investigator) following a previous dose of vaccine.
* (For group 1 only: Criteria for termination of 2nd dose of vaccination) Positive result for SARS-CoV-2 (positive RT-PCR test).
* (For group 1 only: Criteria for termination of 2nd dose of vaccination) The investigator considers inappropriate for the participants to continue participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Incidence, severity, and duration of each solicited (local and systemic) AE. | Within 30 minutes and 7 days after (each dose of) vaccination
Incidence, severity, and duration of each unsolicited AE. | Within 28 days after (each dose of) vaccination
The percentage of participants with abnormal hematology and chemistry laboratory values. | 4 days after (each dose of) vaccination

SECONDARY OUTCOMES:
Geometric Mean Titer (GMT) of SARS-CoV-2 Virus Neutralizing Antibody (VNA) (live virus assay). | Before (each dose of) vaccination, 14 days and 28 days after (each dose of) vaccination
Seroconversion Rate (SCR) of SARS-CoV-2 Virus Neutralizing Antibody (VNA) (live virus assay). | Before (each dose of) vaccination, 14 days and 28 days after (each dose of) vaccination
Geometric Mean Increase (GMI) of SARS-CoV-2 Virus Neutralizing Antibody (VNA) (live virus assay). | Before (each dose of) vaccination, 14 days and 28 days after (each dose of) vaccination
GMT of S-protein specific IgG antibodies (ELISA) | Before (each dose of) vaccination, 14 days and 28 days after (each dose of) vaccination
SCR of S-protein specific IgG antibodies (ELISA) | Before (each dose of) vaccination, 14 days and 28 days after (each dose of) vaccination
GMI of S-protein specific IgG antibodies (ELISA) | Before (each dose of) vaccination, 14 days and 28 days after (each dose of) vaccination
The incidence, severity, and causality of Serious Adverse Events (SAEs) | Within 12 months after (full) vaccination
The incidence, severity, and causality of Adverse Events of Special Interest (AESI) | Within 12 months after (full) vaccination
The incidence, severity, and causality of the occurrence of pregnancy events | Within 12 months after (full) vaccination

OTHER OUTCOMES:
GMT of SARS-CoV-2 VNA (live virus assay). | 3 months and 6 months after (full) vaccination
SCR of SARS-CoV-2 VNA (live virus assay). | 3 months and 6 months after (full) vaccination
GMI of SARS-CoV-2 VNA (live virus assay). | 3 months and 6 months after (full) vaccination
GMT of S-protein specific IgG antibodies (ELISA) | 3 months and 6 months after (full) vaccination
SCR of S-protein specific IgG antibodies (ELISA) | 3 months and 6 months after (full) vaccination
GMI of S-protein specific IgG antibodies (ELISA) | 3 months and 6 months after (full) vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. M. Raza Shah, Principal Investigator — Center for Bioequivalence Studies and Clinical Research